CLINICAL TRIAL: NCT05285475
Title: Effect of Functional Exercises With Water Intake on Sleep Quality and Menstrual Symptoms in Primary Dysmenorrhea
Brief Title: Functional Exercises With Water Intake in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 024433
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Primary Dysmenorrhea
Keywords: Functional exercises, water intake, Menstrual Pain, Sleep
MeSH Terms: conditions — Dysmenorrhea | interventions — Exercise; Drinking

STUDY DESIGN:
Intervention Model Description: There will be two parallel groups in the study.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be kept blind from the group allocation of the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The exercise protocol for this group will be abdominals, pelvic stretching and kegels exercises (PFM) for three days/week lasting about 30 minutes with approximately 1600-1800ml (8-10 glasses) intake of water for 8 weeks (two consecutive menstrual cycles)
  Exercises include:
  Piriformis stretching (5 repetitions×20 seconds) Adductor stretching (5 repetitions×20 seconds) Sit-ups (10 repetitions×3 sets) Bridging (10 repetitions×3 sets) Kegels exercises (10 repetions×3 sets) Pelvic elevation (10 repetitions×3 sets) Pelvic rotation (10 repetitions×3 sets) Cobra pose (5 repetitions×20 seconds)
  Interventions: Other: Exercise and Water Intake
- Group B (No Intervention): The participants in this group will be asked neither to do any exercise nor to change their daily basis routine.

INTERVENTIONS:
Other: Exercise and Water Intake — The exercise protocol for this group will be abdominals, pelvic stretching and kegels exercises (PFM) for three days/week lasting about 30 minutes with approximately 1600-1800ml (8-10 glasses) intake of water for 8 weeks (two consecutive menstrual cycles)
  Exercises include:
  Piriformis stretching (5 repetitions×20 seconds) Adductor stretching (5 repetitions×20 seconds) Sit-ups (10 repetitions×3 sets) Bridging (10 repetitions×3 sets) Kegels exercises (10 repetions×3 sets) Pelvic elevation (10 repetitions×3 sets) Pelvic rotation (10 repetitions×3 sets) Cobra pose (5 repetitions×20 seconds)
  Arms: Group A

SUMMARY:
Dysmenorrhea and its associated symptoms are very common in women. In Pakistan, almost 78% of women report Primary Dysmenorrhea. This will be a randomized controlled trial with two parallel groups. one group will be receiving functional exercises along with water intake and the other will be receiving no interventions.

DETAILED DESCRIPTION:
Mostly in the reproductive years of age women suffers from the Pain of Menstruation which is known as Dysmenorrhea. In Pakistan every other girl is silently suffers from this disease leading to the inefficiency and one of the main cause of school and work absenteeism. This novel study is designed to target the menstrual symptoms of women with functional exercises combine with optimal intake of water. The objective of this study is to determine the effects of functional exercises with water intake on menstrual symptoms and pain in Primary Dysmenorrhea.

This is a Randomized controlled study. Before the study, all the participants will go through baseline evaluation, and then allocated to the groups. The exercise protocol consisting of the combination of exercises with regular intake of water (in bouts) will be informed to them. Females fulfilling the criteria and willing to participate in exercise trial will be recruited in the study. Outcome will be assessed at baseline and post treatment after 8th week.

ELIGIBILITY:
Inclusion Criteria:

* Age group 15-35
* Patients with pain at a severity level of 5 on NPRS during menstruation.
* Primary Dysmenorrhea diagnosis made on WALIDD score
* Patients having regular menstrual cycle

Exclusion Criteria:

* Patients having some previous surgical history
* Patients diagnosed with Secondary Dysmenorrhea
* Abnormal Cognition
* Involved in any regular physical activity for last 6 months

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | changes from Baseline to 8th week
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) is a one-dimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (no pain) to '10' representing the other pain extreme (or "worst pain imaginable"). The intrarater reliability with ICC = 0.67.
Numeric Pain Rating Scale (NPRS) | Post 8 weeks
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) is a one-dimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (no pain) to '10' representing the other pain extreme (or "worst pain imaginable"). The intrarater reliability with ICC = 0.67.
Menstrual Symptom Questionnaire (MSQ) | changes from Baseline to 8th week
  The menstrual symptom questionnaire is a Psychometric test used to determine the menstrual symptoms. The questionnaire consists of 24 items
Menstrual Symptom Questionnaire (MSQ) | post 8th week
  The menstrual symptom questionnaire is a Psychometric test used to determine the menstrual symptoms. The questionnaire consists of 24 items
Pittsburgh Sleep Quality Index (PSQI) | changes from Baseline to 8th week
  The Pittsburg Sleep Quality Index (PSQI) is used to evaluate sleep quality with score ranging from 0 to 21. Higher scores indicate poor sleep quality
Pittsburgh Sleep Quality Index (PSQI) | post 8th week
  The Pittsburg Sleep Quality Index (PSQI) is used to evaluate sleep quality with score ranging from 0 to 21. Higher scores indicate poor sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Behbud Association of Pakistan, Rawalpindi, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirmizigil B, Demiralp C. Effectiveness of functional exercises on pain and sleep quality in patients with primary dysmenorrhea: a randomized clinical trial. Arch Gynecol Obstet. 2020 Jul;302(1):153-163. doi: 10.1007/s00404-020-05579-2. Epub 2020 May 15. PMID 32415471
- [Background] Mahvash N, Eidy A, Mehdi K, Zahra MT, Mani M, Shahla H. The effect of physical activity on primary dysmenorrhea of female university students. World Applied Sciences Journal. 2012;17(10):1246-52.
- [Background] Ortiz MI, Cortes-Marquez SK, Romero-Quezada LC, Murguia-Canovas G, Jaramillo-Diaz AP. Effect of a physiotherapy program in women with primary dysmenorrhea. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:24-9. doi: 10.1016/j.ejogrb.2015.08.008. Epub 2015 Aug 17. PMID 26319652
- [Background] Rakhshaee Z. Effect of three yoga poses (cobra, cat and fish poses) in women with primary dysmenorrhea: a randomized clinical trial. J Pediatr Adolesc Gynecol. 2011 Aug;24(4):192-6. doi: 10.1016/j.jpag.2011.01.059. Epub 2011 Apr 21. PMID 21514190